CLINICAL TRIAL: NCT06557083
Title: The Effects of Practicing Daily Polyvagal Exercises for Four Weeks on Stress in Students of Physical Therapy Measured: a Randomized Controlled Trial
Brief Title: The Effects of Daily Polyvagal Exercises on Stress in Students of Physical Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dominican University New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: DUNY
Record Dates: First submitted 2024-06-25; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Stress; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control, Controlling Stress (Sham Comparator): No intervention will be administered. The control participants will watch a video emphasizing the importance of stress management
  Interventions: Other: No Intervention
- Breathing Exercises (Experimental): The participants in the intervention group will receive a home exercise program (HEP) of Polyvagal breathing exercises. They are instructed to complete these exercises for at least five minutes per day. They are allowed to choose between the three exercises we provide.
  Interventions: Behavioral: Polyvagal Breathing Exercises

INTERVENTIONS:
Behavioral: Polyvagal Breathing Exercises — Breathing exercises provided include, square breathing, modified Qigong breathing, and three step breathing
  Arms: Breathing Exercises
Other: No Intervention — The control group will not perform any intervention.
  Arms: Control, Controlling Stress

SUMMARY:
The purpose of this study is to investigate whether specific breathing exercises can stimulate the polyvagal system and thus decrease stress in healthy students of physical therapy. The hypothesis is that practicing daily polyvagal breathing exercises will result in decreased stress/anxiety in physical therapy students compared to the control group who will not be receiving any intervention.

DETAILED DESCRIPTION:
The study involves healthy physical therapy students of Dominican University New York (DUNY) aged 18-45 who are currently not taking anti-anxiety or anti-depression medications. The independent variable consists of practicing polyvagal breathing exercises over a 30-day period. Only the experimental/breathing group will receive treatment while the control group will not. The dependent variable, stress/anxiety labels, will be measured non-invasively using equipment such as the model number DSI-7 headset to record electroencephalogram (EEG) signals of the brain, which is commonly used in research and considered to be safe. Also, the use of surveys and questionnaires will be utilized.

The DSI-7 headset will be placed on a participant's head in order to utilize the dry sensors to record the electroencephalogram signals of the brain. This headset allows us to read the EEG signals without injecting, inserting, or applying heavy pressure to the participant's head. The participants will be seated during recording of DSI-7 and thus at minimal risk of injury.

Participants will perform three data collections: day one, day fifteen, and day thirty. Participants' brain activity will be measured six times on the day one and day thirty. The first reading, baseline EEG will be recorded while the participant is sitting in a quiet room. They will have their eyes open. The investigators will record their baselines three times for one minute and thirty seconds each. They then will be given three separate seven question timed quizzes via Kahoot in order to induce a small amount of stress. During the quizzes, EEG recordings will be collected. The participant will not receive physical harm nor long term stress. On day fifteen, four EEG recordings will be collected, one at baseline and three during the timed quizzes.

Further, all questionnaires and instructions including the breathing exercises will be given via computer. Each participant in the breathing exercise group will be provided with video instructions on the three breathing exercises and all surveys and questionnaires will be filled out using one laptop to ensure continuity for each participant. The control group will only shown a video with a brief introduction on the ill effects of stress and general tips to relieving stress. However, all participants will receive brain activity readings via EEG.

Participants will be able to withdraw from the study at any given time if they wish to, feel uncomfortable, or experience any adverse effects. The study will be conducted under the supervision of experienced researchers who will follow appropriate safety protocols to minimize any potential risks to participants.

ELIGIBILITY:
Inclusion Criteria:

* Student of physical therapy

Exclusion Criteria:

* Taking medications to treat anxiety or depression

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Stress Levels | 10 minutes
  Utilizing at electroencephalography at baseline, during a short stress induced task (a 7 question timed quiz, performed three times), and after the timed stress inducing task.
  Q-Stats, a program to analyze the raw data, will be utilized to interpret the findings. The data is linearized. The lower the number, the more calm the individual is. (Thus, it is assumed the stress levels are decreased.
Anxiety Levels | 10 minutes
  Utilizing at electroencephalography at baseline, during a short stress induced task (a 7 question timed quiz, performed three times), and after the timed stress inducing task. Q-Stats, a program to analyze the raw data, will be utilized to interpret the findings. The data is linearized. The lower the number, the more calm the individual is. (Thus, it is assumed the anxiety levels are decreased.

SECONDARY OUTCOMES:
10 Item Perceived Stress Scale | 3 minutes
  PSS-10. There are 10 questions. Each question is on a scale of 0 - 4. The scale ranges between 0 and 40. Higher scores are indicate high stress while lower scores indicate low stress.
  Research tool that measures self perceived stress.
7 Item Generalized Anxiety Disorder | 3 minutes
  GAD-7. There are There are 7 questions. Each question is on a scale of 0 - 3. The scale ranges between 0 and 21. Higher scores are indicate severe anxiety while lower scores indicate minimal anxiety.
  Research tool that measures self perceived anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Miscia, Principal Investigator — Dominican University New York; Elise Kang, Principal Investigator — Dominican University New York; Ariane Hasbrouck, Principal Investigator — Dominican University New York
Locations (1):
- Dominican University New York, Orangeburg, New York, United States

IPD SHARING:
Plan to Share IPD: No
Participant information is only accessible by the principal investigators and central contacts.

REFERENCES:
- [Background] Kopplin CS, Rosenthal L. The positive effects of combined breathing techniques and cold exposure on perceived stress: a randomised trial. Curr Psychol. 2022 Oct 7:1-13. doi: 10.1007/s12144-022-03739-y. Online ahead of print. PMID 36248220
- [Background] Magnon V, Dutheil F, Vallet GT. Benefits from one session of deep and slow breathing on vagal tone and anxiety in young and older adults. Sci Rep. 2021 Sep 29;11(1):19267. doi: 10.1038/s41598-021-98736-9. PMID 34588511
- [Background] Porges SW. Orienting in a defensive world: mammalian modifications of our evolutionary heritage. A Polyvagal Theory. Psychophysiology. 1995 Jul;32(4):301-18. doi: 10.1111/j.1469-8986.1995.tb01213.x. PMID 7652107
- [Background] Aranberri-Ruiz A, Aritzeta A, Olarza A, Soroa G, Mindeguia R. Reducing Anxiety and Social Stress in Primary Education: A Breath-Focused Heart Rate Variability Biofeedback Intervention. Int J Environ Res Public Health. 2022 Aug 17;19(16):10181. doi: 10.3390/ijerph191610181. PMID 36011817